CLINICAL TRIAL: NCT02091986
Title: A Phase 3, 12-Week, Double-Blind, Randomized, Parallel-Group, Multicenter Study Investigating the Efficacy and Safety of Symbicort pMDI 80/2.25 μg, 2 Actuations Twice Daily, and Symbicort pMDI 80/4.5 μg, 2 Actuations Twice Daily, Compared With Budesonide pMDI 80 μg, 2 Actuations Twice Daily, in Children Ages 6 to <12 Years With Asthma
Brief Title: A 12-Week Study in Asthmatic Children Ages 6 to <12 Years, Investigating the Efficacy and Safety of Symbicort pMDI 80/2.25 μg and Symbicort pMDI 80/4.5 μg, Compared With Budesonide pMDI 80 μg
Acronym: CHASE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589GC00003
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: asthma, children, budesonide pMDI
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Symbicort pMDI 80/2.25 µg (Active Comparator): Budesonide/formoterol pMDI 80/2.25 µg, 2 acuations twice daily
  Interventions: Drug: Symbicort pMDI
- Symbicort pMDI 80/4.5µg (Active Comparator): Budesonide/formoterol pMDI 80/4.5µg, 2 acuations twice daily
  Interventions: Drug: Symbicort pMDI
- Budesonide pMDI (Active Comparator): Budesonide pMDI 80µg, 2 acuations twice daily
  Interventions: Other: Budesonide pMDI

INTERVENTIONS:
Drug: Symbicort pMDI — Budesonide/formoterol pMDI 80/2.25 µg, 2 acuations twice daily
  Arms: Symbicort pMDI 80/2.25 µg
Drug: Symbicort pMDI — Budesonide/formoterol pMDI 80/4.5µg, 2 acuations twice daily
  Arms: Symbicort pMDI 80/4.5µg
Other: Budesonide pMDI — Budesonide pMDI 80µg, 2 acuations twice daily
  Other Names: Active comparator
  Arms: Budesonide pMDI

SUMMARY:
The purpose is to investigate the Efficacy and Safety of Symbicort pMDI 80/2.25 μg and Symbicort pMDI 80/4.5 μg, Compared with Budesonide pMDI 80 μg, 2 Actuations Twice Daily, in Children Ages 6 to <12 Years with Asthma during 12 weeks.

DETAILED DESCRIPTION:
A Phase 3, 12-Week, Double-Blind, Randomized, Parallel-Group, Multicenter Study Investigating the Efficacy and Safety of Symbicort pMDI 80/2.25 μg, 2 Actuations Twice Daily, and Symbicort pMDI 80/4.5 μg, 2 Actuations Twice Daily, Compared with Budesonide pMDI 80 μg, 2 Actuations Twice Daily, in Children Ages 6 to <12 Years with Asthma

ELIGIBILITY:
Inclusion Criteria:

* Has a documented clinical diagnosis of asthma defined by the ATS for at least 6 months prior to Visit 2
* Have a morning pre-bronchodilator clinic FEV1 measured at least 6 hours after the last dose of inhaled SABA and at least 48 hours after last dose of inhaled LABA of 60% to 100% of predicted normal
* Demonstrated reversibility of clinic FEV1 of ≥12% from pre -albuterol/salbutamol level within 15 to 30 minutes after administration of a standard dose of albuterol/salbutamol.

Exclusion Criteria:

* Have been hospitalized at least once or required emergency treatment more than once for an asthma-related condition during the 6 months prior to Visit 1
* Have required treatment with systemic corticosteroids (eg, oral, parenteral, or rectal) for any reason within the 6 weeks prior to Visit 1

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 882 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Pearlman, MD, Principal Investigator — Colorado Allergy Asthma Centers, PC, US; Carin Jorup, MD, Study Director — AstraZeneca Mölndal, Sweden
Locations (70):
- United States (59):
  - Research Site, Hoover, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Ontario, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Fort Walton Beach, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Williston, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Lenexa, Kansas
  - Research Site, Waldorf, Maryland
  - Research Site, Plymouth, Minnesota
  - Research Site, Bellevue, Nebraska
  - Research Site, Verona, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rockville Centre, New York
  - Research Site, Watertown, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Gresham, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Upland, Pennsylvania
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Allen, Texas
  - Research Site, Baytown, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerville, Texas
  - Research Site, Richmond, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Murray, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Washington, Washington
- Mexico (3):
  - Research Site, Cuautitlán Izcalli
  - Research Site, México
  - Research Site, Monterrey
- Panama (2):
  - Research Site, David Chiriqui
  - Research Site, Panama City
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Poprad
  - Research Site, Prešov

REFERENCES:
- [Derived] Pearlman DS, Eckerwall G, McLaren J, Lamarca R, Puu M, Gilbert I, Jorup C, Sandin K, Lanz MJ. Efficacy and safety of budesonide/formoterol pMDI vs budesonide pMDI in asthmatic children (6-<12 years). Ann Allergy Asthma Immunol. 2017 Apr;118(4):489-499.e1. doi: 10.1016/j.anai.2017.01.020. Epub 2017 Mar 1. PMID 28256307

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the protocol section denotes the number of patients screened into the trial. Out of these 882 patients screened, 279 patients were randomized into the trial. This explains the discrepancy in patient number.
Groups:
- Symbicort pMDI 80/4.5 ug; Symbicort pMDI 80/2.25 ug: Symbicort pMDI 80/4.5 ug x 2 BID
- Budesonide pMDI 80 ug: Budesonide pMDI 80 ug x 2 BID
Period: Overall Study
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Started | 92 | 95 | 92
Completed | 85 | 84 | 84
Not Completed | 7 | 11 | 8
Not completed — 7 rand in error 1 patient decision | 2 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 3
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All patients randomized, defined as having a randomization code recorded on the demography case report form (CRF)
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug | Total
Number analyzed (Participants) | 92 | 95 | 92 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (1.6) | 9 (1.6) | 9 (1.4) | 9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 37 | 113
  Male | 50 | 61 | 55 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 36 | 32 | 106
  Not Hispanic or Latino | 54 | 59 | 60 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 3 | 8
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 24 | 26 | 26 | 76
  White | 61 | 60 | 53 | 174
  More than one race | 4 | 4 | 7 | 15
  Unknown or Not Reported | 0 | 2 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 38 (12.9) | 38 (12.9) | 40 (13.6) | 39 (13.1)
Height [Mean (Standard Deviation); unit: cm] | 139 (11.1) | 138 (10.9) | 141 (10.5) | 139 (10.8)
Duration of asthma [Mean (Standard Deviation); unit: years] | 5.8 (3.0) | 5.9 (3.2) | 6.2 (3.1) | 5.9 (3.1)
FEV1 at randomisation [Mean (Standard Deviation); unit: Liters] | 1.58 (0.42) | 1.57 (0.33) | 1.62 (0.36) | 1.59 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in 1h Post-dose FEV1
Description: 1h post-dose FEV1 is defined as the 1-hour post-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: All patients randomized who:
  * received at least one dose of study medication;
  * the patient contributed data for at least one efficacy endpoint.
  Patients accounted for according to the treatment to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Symbicort pMDI 80/2.25 ug: Symbicort pMDI 80/2.25 ug x 2 BID
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 90 | 93 | 90
Liters | 0.28 [0.22 to 0.34] | 0.24 [0.18 to 0.31] | 0.17 [0.10 to 0.23]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Baseline FEV1, Treatment group, Region, Age were all included as explanatory variables in the linear predictor
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis; Baseline FEV1, Treatment group, Region, Age were all included as explanatory variables in the linear predictor
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis; Baseline FEV1, Treatment group, Region, Age were all included as explanatory variables in the linear predictor

2. Secondary Outcome: Change From Baseline to Week 12 in 1h Post-dose PEF
Description: 1h post-dose PEF is defined as the 1-hour post-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 93 | 90
Liters per minute | 57.04 [46.12 to 67.97] | 41.14 [30.26 to 52.01] | 31.57 [20.78 to 42.36]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Baseline lung function assessment, Treatment group, Region, Age were all included as explanatory variables in the linear predictor
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.195, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline to Week 12 in 1h Post-dose FEF25-75
Description: 1h post-dose FEF25-75 is defined as the 1-hour post-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per second
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 93 | 90
Liters per second | 0.55 [0.43 to 0.67] | 0.47 [0.35 to 0.59] | 0.23 [0.11 to 0.35]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.326, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline to Week 12 in 1h Post-dose FVC
Description: 1h post-dose FVC is defined as the 1-hour post-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 93 | 90
Liters | 0.22 [0.15 to 0.30] | 0.16 [0.09 to 0.23] | 0.17 [0.10 to 0.24]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.276, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.759, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.165, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline to Week 12 in Pre-dose FEV1
Description: Pre-dose FEV1 is defined as the pre-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 92 | 89
Liters | 0.11 [0.04 to 0.17] | 0.10 [0.03 to 0.16] | 0.09 [0.03 to 0.15]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.724, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.909, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.811, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline to Week 12 in Pre-dose PEF
Description: Pre-dose PEF is defined as the pre-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 92 | 89
Liters per minute | 27.73 [16.37 to 39.08] | 15.86 [4.39 to 27.33] | 16.01 [4.50 to 27.52]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.134, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.985, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 12 in Pre-dose FEF25-75
Description: Pre-dose FEF25-75 is defined as the pre-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 92 | 89
Liters per minute | 0.12 [0.01 to 0.24] | 0.13 [0.01 to 0.25] | 0.09 [-0.03 to 0.21]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.684, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.621, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: Change From Baseline to Week 12 in Pre-dose FVC
Description: Pre-dose FVC is defined as the pre-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 89 | 92 | 89
Liters | 0.11 [0.03 to 0.18] | 0.11 [0.04 to 0.19] | 0.13 [0.05 to 0.20]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.664, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.747, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.913, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

9. Secondary Outcome: Change From Baseline to Week 12 in 15 Min Post-dose FEV1
Description: 15 min Post-dose FEV1 is defined as the 15 min post-dose measurement taken at Week 12 minus the pre dose measurement taken at randomization for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 79 | 78 | 80
Liters | 0.25 [0.18 to 0.31] | 0.19 [0.12 to 0.25] | 0.15 [0.08 to 0.21]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.015, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.342, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.138, ANCOVA; [statistical method as in outcome 2, analysis 1]

10. Secondary Outcome: Change From Baseline to End of Study Average in Total Asthma Symptoms
Description: End of study average is defined as the average of available records from 7 days before up to and including the day prior to withdrawal from study or Week 12, minus the baseline measurement at randomization, for patients who remain in the study (irrespective of whether IP has been discontinued).
  Patient to record his/her asthma symptom score twice daily. The following rating scales are to be used: 0 = None; no symptoms of asthma
  1. = Mild symptoms; awareness of asthma symptoms and/or signs that are easily tolerated
  2. = Moderate symptoms, asthma symptoms with some discomfort, causing some interference with daily activities or sleep
  3. = Severe symptoms; incapacitating asthma symptoms and/or signs, with inability to perform daily activities or to sleep
  Total asthma symptom score is derived as the sum of the daytime score plus the score from the previous nighttime, ie possible range (0 to 6).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 70 | 72 | 73
units on a scale | -0.5 (0.73) | -0.6 (0.73) | -0.4 (0.55)

11. Secondary Outcome: Change From Baseline to End of Study Average in % of Night Time Awakenings Due to Asthma Symptoms
Description: End of study average is defined as the percentage of nighttime awakenings due to asthma symptoms from 6 days before up to and additionally including the morning of withdrawal from study or Week 12, minus the baseline measurement at randomization, for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of nighttime awakenings
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 79 | 85 | 82
Percentage of nighttime awakenings | -14.0 (29.15) | -17.3 (33.16) | -13.0 (21.87)

12. Secondary Outcome: Change From Baseline to End of Study Average in Total Daily Reliever Medication
Description: End of study average is defined as the average of available records from 7 days before up to and including the day prior to withdrawal from study or Week 12, minus the baseline measurement at randomization, for patients who remain in the study (irrespective of whether IP has been discontinued).
Time Frame: Week 0 (baseline), Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of reliever medication use
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 70 | 72 | 73
Number of reliever medication use | -0.7 (1.75) | -1.1 (2.37) | -0.7 (1.37)

13. Secondary Outcome: Change From Baseline to Study Period Average in Overall PAQLQ Score
Description: Study period average is defined as the average of the post-baseline values during the study taken after first dose of investigational product up to and including withdrawal from study or Week 12, minus the baseline assessment at randomization, for patients who remain in the study (irrespective of whether IP has been discontinued).
  The PAQLQ(S) is a 23-item patient-reported questionnaire, each one reported on a 7-point scale (e.g. 1 = extremely bothered/all of the time; 7 = not bothered/none of the time). The PAQLQ(S) generates an overall score, as well as 3 domain scores: activity limitations (5 items), symptoms (10 items) and emotional function (8 items). The overall score will be calculated as the mean of the responses to each of the 23 questions (ie the range of 1-7, where higher scores indicate better quality of life). If any of the domain scores are missing, no total score will be calculated.
Time Frame: Week 0 (baseline), week 4, week 8, week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: unit on a scale
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 79 | 80 | 82
unit on a scale | 0.46 [0.30 to 0.62] | 0.53 [0.38 to 0.69] | 0.62 [0.47 to 0.78]
Statistical Analysis 1: Comparison: Symbicort pMDI 80/4.5 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.098, ANCOVA; The explanatory variables included in the model are: treatment group, baseline overall PAQLQ(S) score, region and age group
Statistical Analysis 2: Comparison: Symbicort pMDI 80/2.25 ug vs Budesonide pMDI 80 ug; Test type: Superiority or Other; p = 0.367, ANCOVA; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Symbicort pMDI 80/4.5 ug vs Symbicort pMDI 80/2.25 ug; Test type: Superiority or Other; p = 0.449, ANCOVA; [statistical method as in outcome 13, analysis 1]

14. Secondary Outcome: Number of Patients With an Asthma Exacerbation During Study
Description: Number of patients that experienced an asthma exacerbation that required either emergency room treatment, hospitalization, systemic steroids, or an increase in, or additional asthma maintenance medication, during the study.
Time Frame: Week 0 (baseline) up to Week 12
Population: All patients randomized who:
  * received at least one dose of study medication;
  * data collected after randomisation. Patients accounted for according to the treatment they actually received.
Measure: Number; unit: Partcicipants
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Number analyzed (Participants) | 90 | 93 | 90
Partcicipants | 9 | 12 | 12

ADVERSE EVENTS:
Time Frame: Week 0 (baseline) up to 12 weeks
Description: Serious Adverse Events Table, Other Adverse Events Table based on all of patients rand who :
  * received at least 1 dose of study meds;
  * data were collected after randomization. No of part provided in the Participant Flow Module based on all patients randomized.
Arm/Group | Symbicort pMDI 80/4.5 ug | Symbicort pMDI 80/2.25 ug | Budesonide pMDI 80 ug
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/93 | 2/90
Other Adverse Events (participants affected / at risk) | 42/90 | 41/93 | 40/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort pMDI 80/4.5 ug (N=90) | Symbicort pMDI 80/2.25 ug (N=93) | Budesonide pMDI 80 ug (N=90)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort pMDI 80/4.5 ug (N=90) | Symbicort pMDI 80/2.25 ug (N=93) | Budesonide pMDI 80 ug (N=90)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 10
Upper respiratory tract infection (Infections and infestations) | 9 | 12 | 4
Pyrexia (General disorders) | 4 | 4 | 4
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Pharyngitis (Infections and infestations) | 5 | 3 | 1
Headache (Nervous system disorders) | 4 | 4 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 1
Influenza (Infections and infestations) | 1 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 2
Rhinitis (Infections and infestations) | 3 | 2 | 2
Viral upper respiratory tract (Infections and infestations) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No